CLINICAL TRIAL: NCT03323190
Title: An Educational Intervention to Improve Disease Management Knowledge of Hospitalized Patients With COPD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn due to low feasibility.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15121607-IRB04
Record Dates: First submitted 2017-02-10; First posted 2017-10-26 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Chronic Obstructive Pulmonary Disease; Patient Education; Inpatients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inpatient COPD patient (Experimental): All COPD patients meeting the inclusion criteria of this study will be exposed to inpatient COPD education and tested at a later date to determine if knowledge on COPD was gained.
  Interventions: Behavioral: Inpatient COPD education

INTERVENTIONS:
Behavioral: Inpatient COPD education

SUMMARY:
The objective of this study is to determine if inpatient COPD education would result in improved patient knowledge of COPD.

DETAILED DESCRIPTION:
A prospective cohort study utilizing a pre-test/post-test design will be used to test a COPD education intervention on a convenience sample of 30 patients with a diagnosis of COPD. Study participants will complete the Chronic Obstructive Pulmonary Disease questionnaire (COPD-Q) to assess their COPD knowledge. Next, a respiratory therapist will provide the first scripted COPD education session. The patient will complete the COPD-Q 24 hours and 30 days post-discharge. Demographic data, smoking status, pack-years, COPD spirometry grade, COPD symptom and exacerbation grade, previous hospital admissions, support system for managing COPD, attendance at previous formal education for COPD, current and home medications, pulmonary function test (PFT) results, vaccinations, and level of education data will be collected. Data related to patient recruitment will also be collected. Means and standard deviation will be reported for interval data. Total frequency and percentages will be reported for nominal data, and median and 25th and 75th percentile will be reported for COPD severity. Repeated measures ANOVA (p< 0.05) will be used to evaluate if an inpatient COPD self-management intervention can increase the patient's knowledge of COPD after 24 hours and again at 30 days after the initial education session.

This study is expected to show that an inpatient education of COPD can increase the patient's COPD knowledge prior to discharge and that it will be retained for at least one month post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* History of COPD
* Spirometry confirmation of COPD either from chart or bedside spirometry i. FEV1(forced expiatory volume in 1 second)/FVC (forced vital capacity) <70% ii. FEV1 < 80% predicted
* Willingness to participate
* English-speaking
* Working phone

Exclusion Criteria:

* Cognitively impaired (including sedation)
* Intubated
* Non-English-speaking
* Receiving palliative or hospice service
* Enrolled in any other educational research s

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Gained knowledge | 1 year
  Change from baseline on the Chronic Obstructive Pulmonary Disease Questionnaire (COPD-Q).

SECONDARY OUTCOMES:
Pulmonary rehab enrollment | 1 year
  Number of subjects that have enrolled in pulmonary rehab.

CONTACTS AND LOCATIONS:
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sayiner A, Alzaabi A, Obeidat NM, Nejjari C, Beji M, Uzaslan E, Nafti S, Khan JA, Tageldin MA, Idrees M, Rashid N, El Hasnaoui A; BREATHE Study Group. Attitudes and beliefs about COPD: data from the BREATHE study. Respir Med. 2012 Dec;106 Suppl 2:S60-74. doi: 10.1016/S0954-6111(12)70015-X. PMID 23290705
- [Background] Cramm JM, Nieboer AP. The relationship between self-management abilities, quality of chronic care delivery, and wellbeing among patients with chronic obstructive pulmonary disease in The Netherlands. Int J Chron Obstruct Pulmon Dis. 2013;8:209-14. doi: 10.2147/COPD.S42667. Epub 2013 Apr 26. PMID 23641152
- [Background] Zwar NA, Hermiz O, Comino E, Middleton S, Vagholkar S, Xuan W, Wilson SF, Marks GB. Care of patients with a diagnosis of chronic obstructive pulmonary disease: a cluster randomised controlled trial. Med J Aust. 2012 Oct 1;197(7):394-8. doi: 10.5694/mja12.10813. PMID 23025736
- [Background] Maples P, Franks A, Ray S, Stevens AB, Wallace LS. Development and validation of a low-literacy Chronic Obstructive Pulmonary Disease knowledge Questionnaire (COPD-Q). Patient Educ Couns. 2010 Oct;81(1):19-22. doi: 10.1016/j.pec.2009.11.020. Epub 2009 Dec 30. PMID 20044232
- [Background] Messenger RW. Reducing chronic obstructive pulmonary disease readmissions: the role of the durable medical equipment provider. Prof Case Manag. 2012 May-Jun;17(3):109-14; quiz 115-6. doi: 10.1097/NCM.0b013e31823ba2b8. PMID 22488339
- [Background] Cooney A, Mee L, Casey D, Murphy K, Kirwan C, Burke E, Conway Y, Healy D, Mooney B, Murphy J; PRINCE Team. Life with chronic obstructive pulmonary disease: striving for 'controlled co-existence'. J Clin Nurs. 2013 Apr;22(7-8):986-95. doi: 10.1111/j.1365-2702.2012.04285.x. Epub 2013 Jan 2. PMID 23279604
- [Background] Taylor SJ, Candy B, Bryar RM, Ramsay J, Vrijhoef HJ, Esmond G, Wedzicha JA, Griffiths CJ. Effectiveness of innovations in nurse led chronic disease management for patients with chronic obstructive pulmonary disease: systematic review of evidence. BMJ. 2005 Sep 3;331(7515):485. doi: 10.1136/bmj.38512.664167.8F. Epub 2005 Aug 10. PMID 16093253
- [Background] Adis Medical Writers. (2013). Managing coexistent asthma and chronic obstructive pulmonary disease in older populations is challenging. Drugs & Therapy Perspectives, 29, 141-144.
- [Background] Jones PW, Adamek L, Nadeau G, Banik N. Comparisons of health status scores with MRC grades in COPD: implications for the GOLD 2011 classification. Eur Respir J. 2013 Sep;42(3):647-54. doi: 10.1183/09031936.00125612. Epub 2012 Dec 20. PMID 23258783
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Duley L, Antman K, Arena J, Avezum A, Blumenthal M, Bosch J, Chrolavicius S, Li T, Ounpuu S, Perez AC, Sleight P, Svard R, Temple R, Tsouderous Y, Yunis C, Yusuf S. Specific barriers to the conduct of randomized trials. Clin Trials. 2008;5(1):40-8. doi: 10.1177/1740774507087704. PMID 18283079
- [Background] Lawlor M, Kealy S, Agnew M, Korn B, Quinn J, Cassidy C, Silke B, O'Connell F, O'Donnell R. Early discharge care with ongoing follow-up support may reduce hospital readmissions in COPD. Int J Chron Obstruct Pulmon Dis. 2009;4:55-60. Epub 2009 Apr 15. PMID 19436695